CLINICAL TRIAL: NCT01633437
Title: A Phase I, Multiple-Dose, Randomized, Double-Blind, Oral Tyramine Pressor Response Study Comparing CX157 Tablets to Placebo in Healthy Male Volunteers
Brief Title: Oral Tyramine Pressor Response Study of CX157 Tablets in Healthy Male Volunteers
Acronym: CX157-112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CeNeRx BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CX157-112
Record Dates: First submitted 2012-06-28; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Major Depressive Disorder
Keywords: tyramine; MAOI; cheese effect; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — CX157

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Other: Placebo
- CX157 (Experimental): CX157 is a reversible monoamine oxidase inhibitor (RIMA) in Phase II development for the treatment of depression.
  Interventions: Drug: CX157

INTERVENTIONS:
Drug: CX157 — CX157 Modified Release Tablet 125 mg administered twice per day on study days 4-11 and in the morning of study day 12.
  Arms: CX157
Other: Placebo — Placebo administered twice per day on study days 4-11 and in the morning of day 12.
  Arms: Sugar pill

SUMMARY:
The objectives of this study were to examine the cardiovascular sensitivity to oral tyramine after establishment of steady state with CX157 Modified Release (MR) Tablets, 125 mg administered twice per day (BID) in healthy volunteers compared to placebo; and to investigate the general safety, tolerability and pharmacokinetic profile of CX157 tablets at steady state compared to placebo.

DETAILED DESCRIPTION:
Methodology: The trial was a Phase 1, single center, DB, three-period study of cardiovascular safety following oral administration of encapsulated tyramine prior to treatment with double-blind (DB) study drug (CX157 Modified Release Tablets, 125 mg administered twice per day (BID) or matching placebo administered BID) and the administration of tyramine in yogurt along with a standard meal during the DB study treatment administration, after CX157 reached steady state.

Prior to treatment with DB study treatment, baseline cardiovascular sensitivity to oral tyramine administered in a fasting state was established in 15 subjects during Period 1 Days 1-3. Following completion of Period 1, the study's 12 subjects were randomized to CX157 (10 subjects) or placebo (2 subjects) and treated for six consecutive days (Days 4-9) to reach steady state. Subjects continued their DB study treatment in Period 3 (Days 10-12); however, during this period tyramine was administered to subjects in the fed state on Day 10 (tyramine 20 mg), Day 11 (tyramine 40 mg) and Day 12 (tyramine 80 mg).

The tyramine pressor dose (minimum dose of tyramine necessary to achieve endpoint) for Period 1 was established through a series of three tyramine challenges (24 hours apart) with tyramine doses based upon a predetermined paradigm. During Period 1, untreated fasting subjects received an initial tyramine challenge dose of 400 mg and were monitored for SBP endpoint changes (SBP increase of ≥30 mmHg on three consecutive occasions at least five minutes apart over a 10-minute (i.e., TYR303). If pressor endpoint was achieved, the tyramine challenge dose administered on Period 1 Day 2 was reduced to 200 mg. However, if endpoint was not achieved, the tyramine challenge dose was raised on Period 1 Day 2 to 600 mg. This dose escalation/reduction paradigm was repeated on Period 1 Day 3 based upon the results of Period 1 Day 2 in order to establish the tyramine pressor dose during that period.

During Period 2 (Days 4-9) subjects were treated with CX157 or placebo twice daily to reach the steady state. On Day 8 of Period 2, single-blind yogurt without tyramine was administered with lunch to familiarize subjects and the clinic staff with the procedures for Period 3.

The tyramine challenges for Period 3 Days 10 - 12 began after six consecutive days of treatment with CX157 or placebo twice daily. The tyramine doses for Period 3 were 20, 40, and 80 mg (24 hours apart). The endpoint for Period 3 was the same as described above for Period 1, reaching of the pressor endpoint (i.e., TYR303).

The study planned for 12 healthy male volunteer subjects to be randomized at Period 2. Ten (10) subjects were to be randomized to CX157 MR Tablets, 125 mg and 2 to matching placebo. Approximately 15 subjects were to enter Period 1 in order to ensure randomization of 12 subjects to Period 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 to 50 years of age, inclusive.
2. In good general health as ascertained by not clinically significant physical examination (PE) including measurement of vital signs, medical history, clinical laboratory studies, and 12-lead electrocardiogram (ECG).
3. Body Mass Index (BMI) ≥22 and ≤30 kg/m2.
4. Agree to abstain from consuming either alcohol-containing or caffeine-containing beverages and to adhere to the dietary restrictions.

Exclusion Criteria:

1. Presence of a significant acute or chronic medical disorder.
2. The mean of three consecutive semi-recumbent SBP and diastolic blood pressure (DBP) readings taken five minutes apart over a 10-minute period at Screening and Day -1 exceeds 140 mmHg and 90 mmHg, respectively, and/or is not stable (semi-recumbent SBP exceeds a maximum range of 10 mmHg between the lowest and highest value).
3. The mean of three consecutive semi-recumbent SBP and DBP readings taken five minutes apart over a 10-minute period at Screening and Day -1 is <90 mmHg and 60 mmHg, respectively.
4. Has the requirement for or use of any prescription medications within 35 days of study initiation or anticipates use of any psychoactive medication during the study.
5. Has taken an monoamine oxidase inhibitor (MAOI) within 90 days preceding Period 1, Day 1 of the study.
6. Has requirement for any medication contraindicated for use with an MAOI.
7. Use of any over-the-counter (OTC) medication within 14 days of study drug.
8. History of substance abuse or dependence, including alcohol abuse as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria, within the past 12 months.
9. Use of tobacco products or any nicotine-containing products (e.g., gum, patch) currently or within the prior 6 months.
10. Subject is unwilling to stop consumption of alcohol or caffeine/xanthine-containing drinks or foods within 72 hours of dosing of Day 1 (including any type of wines, caffeinated or decaffeinated herbal tea, grapefruit products (e.g., fresh, canned, or frozen), Seville oranges and pomelos).
11. Subjects with known adverse events associated with ingestion of tyramine-containing food.
12. Subjects with contraindications to administration of adrenergic receptor antagonists such as labetalol (e.g., asthma, obstructive airway disease, severe bradycardia, diabetes).
13. Abnormal screening medical/physical examination, unless the abnormality is considered unlikely to be affected by study participation, or to confound interpretation of safety data.
14. A clinically significant clinical laboratory or ECG abnormality at screening; includes any of the following:

    1. Aspartate aminotransferase (AST/SGOT) >2.0 x the upper limit of normal (ULN),
    2. Alanine aminotransferase (ALT/SGPT) >2.0 x the ULN,
    3. Alkaline phosphatase (ALP) >2.0 x the ULN,
    4. Total bilirubin >1.5 x the ULN,
    5. Serum creatinine >1.5 x the ULN, and
    6. Blood urea nitrogen (BUN) >1.5 x the ULN.
15. Anticipates elective surgery requiring general anesthesia for at least 10 days following the end of study.
16. Test positive for: Cannabinoids, cocaine, amphetamines, barbiturates, opiates or benzodiazepines, cotinine, alcohol use, hepatitis B or C, or human immunodeficiency virus (HIV).
17. Participation in a clinical investigation within the last 60 days.
18. Previous participation in a prior study of CX157.
19. Any other condition which, in the investigator's opinion, may place the subject at greater than normal risk of developing complications.
20. Donated any blood product (one pint or greater) within the previous 8 weeks.
21. Planning to donate any blood product within 8 weeks of end of study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) | 4 hours post dose on study Days 10, 11, 12
  SBP was measured every 5 minutes for the first two hours and every 15 minutes for the next two hours post tyramine ingestion on study Days 10 (20 mg tyramine), 11 (40 mg tyramine), and 12 (80 mg tyramine).

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability of CX157. | Study Days 4-12 (during the DB study drug administration)
  Adverse events were collected during the study.
Cmax, Cmin, Tmax | Study Days 6-12
  The full pharmacokinetic (PK) profile was obtained after the morning dose on Day 9. In addition, trough blood samples were obtained before the morning and evening doses on study Days 6, 7, and 8; and before the morning dose on Days 10, 11 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: William Gerson, D.O., Principal Investigator — Comprehensive Phase One
Locations (1):
- Comprehensive Phase One, Miramar, Florida, United States